CLINICAL TRIAL: NCT04576312
Title: Phase 1 Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Assess the Safety of Ascending Doses of UNI911 INHALATION in Healthy Volunteers in Preparation for Evaluation in Adults With COVID-19
Brief Title: Safety of Ascending Doses of Niclosamide (UNI911 INHALATION) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: UNI911-101; 2020-002049-40 (EudraCT Number)
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Single dose of UNI911 inhalation (4 mL 0.1% ~ 3,4 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg)
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%; Drug: Placebo
- Cohort 2 (Experimental): Single dose of UNI911 inhalation (1 mL 1% ~ 8,4 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg)
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%; Drug: Placebo
- Cohort 3 (Experimental): Single dose of UNI911 inhalation (3 mL 1% ~ 25,2 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg)
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%; Drug: Placebo
- Cohort 4 (Experimental): Single dose of UNI911 inhalation (6 mL 1% ~ 50,4 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg)
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%; Drug: Placebo
- Cohort 5 (Experimental): UNI911 inhalation (6 mL 1% ~ 50,4 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg) BID for 2,5 days.
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%; Drug: Placebo
- Cohort 6 (Experimental): UNI911 inhalation (1 mL 1% ~ 8,4 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg) BID for 6,5 days.
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%
- Cohort 7 (Experimental): UNI911 inhalation (3 mL 1% ~ 25,2 mg) and intranasal spray (2 x 150 µL, 1% ~ 2,5 mg) BID for 6,5 days.
  Interventions: Drug: UNI911 inhalation 1% and intranasal spray 1%
- Placebo (applicable for cohorts 1-5) (Placebo Comparator): Placebo, administered in a double-blinded fashion (except for the first subjects of cohorts 1-4) at the same dose and frequency as UNI911 inhalation and intranasal spray.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UNI911 inhalation 1% and intranasal spray 1% — Niclosamide is a broad spectrum, host tageting antiviral that inhibits viral replication (by neutralizing endosomal pH) and increases viral clearance (by increasing the autophagic flux). The niclosamide 1% solution is administered as inhalation by nebulization and intranasal by a nasal spray.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7
Drug: Placebo — The placebo formulation contains the vehicle. The solution is administered in the same way as the active drug. Placebo was only administered for cohorts 1-5.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Placebo (applicable for cohorts 1-5)

SUMMARY:
This is a Phase 1 Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Assess the Safety of Ascending Doses of UNI911 INHALATION in Healthy Volunteers in Preparation for Evaluation in Adults with COVID-19

DETAILED DESCRIPTION:
This is a Phase 1 Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Assess the Safety of Ascending Doses of UNI911 INHALATION in Healthy Volunteers in Preparation for Evaluation in Adults with COVID-19

64 subjects will be sequentially enrolled to receive dosage of UNI911 INHALATION or placebo. 4 sentinel subjects (one per cohort 1, 2 ,3 and 4 ) will be treated in an open-label manner to confirm the safety of each dose sequentially. 40 subjects will be randomly assigned (3:1) to either active or placebo. For the last 2 cohorts, a total of 20 healthy volunteers will be enrolled to receive multiple doses of UNI911 INHALATION.

ELIGIBILITY:
Inclusion Criteria (main ones):

1. Signed Informed Consent Form (ICF)
2. Male or non-pregnant and non-lactating female who is abstinent or agrees to use effective contraceptive methods throughout the course of the study. Females must have a negative urine beta-human chorionic gonadotropin hormone (hCG) pregnancy test prior to dosing. (Women who are postmenopausal or who had tubal ligation/hysterectomy do not need to have a pregnancy test done and do not need to agree to use contraception.)
3. ECG without clinically significant abnormalities (including QTcF < 450 ms)
4. Age ≥ 18 and < 65 years at the time of signing ICF
5. Normally active and in good health by medical history and physical examination
6. Minimum 80% of predicted lung function, including FEV1 after beta2-agonist, TLC, DCO, and CPET with pulse oximetry
7. Chest X-ray without clinically significant abnormalities

Exclusion Criteria (main ones):

1. Enrollment in an UNI911 study in the previous 6 months
2. Clinically significant allergy (as judged by the investigator) or history of significant adverse reaction to niclosamide or related compounds, to any of the excipients used.
3. Underlying condition that may interfere with inhalation of the IP
4. Current acute or chronic condition (incl. COPD, asthma, or other severe respiratory disease, CV disease, diabetes mellitus, obesity, malignant and autoimmune diseases) unless considered clinically irrelevant and stable by the investigator
5. Renal impairment (eGFR < 60 mL/min/1.73m2) or hepatic impairment (as judged by the investigator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Assess safety of UNI911 INHALATION in healthy volunteers: AE frequency | Up to Day 6
  AE frequency in each cohort and treatment group

OTHER OUTCOMES:
Pharmacokinetic Parameters: Cmax | Up to Day 4 of participant treatment
  Maximum concentration of active drug molecules in blood (Cmax)
Pharmacokinetic Parameters: Tmax | Up to Day 4 of participant treatment
  Time to reach maximum level (Tmax)
Pharmacokinetic Parameters: AUC | Up to Day 4 of participant treatment
  Area Under the Curve of drug level in blood versus time (AUC)
Pharmacokinetic Parameters: Half life | Up to Day 4 of participant treatment
  Half life

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonne, MD, DMSci, Principal Investigator — Dantrials Aps
Locations (1):
- DanTrials ApS, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No